CLINICAL TRIAL: NCT04288427
Title: 5-Alpha Reductase 2 as a Marker of Resistance to 5ARI Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Aria F. Olumi, MD, Principal Investigator; Chief of Urologic Surgery at Beth Israel Deaconess Medical Center; Janet & William DeWolf Professor of Surgery/Urology at Harvard Medical School; American Urological Association Chair of Research, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020P000202; R01DK124502 (NIH)
Record Dates: First submitted 2020-02-10; First posted 2020-02-28 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Benign Prostatic Hyperplasia; Prostate Hyperplasia; Prostate Disease; Prostate Hypertrophy; Prostate Pain; Lower Urinary Tract Symptoms; Urinary Obstruction; Urinary Tract Disease
Keywords: Finasteride; 5 Alpha Reductase
MeSH Terms: conditions — Prostatic Hyperplasia; Prostatic Diseases; Lower Urinary Tract Symptoms; Urologic Diseases | interventions — Finasteride

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Finasteride Treatment (Experimental): Patients who are eligible will be given 5ARI therapy, Finasteride, for medical management of Benign Prostatic Hyperplasia (BPH) symptoms. Only patients with lower urinary tract symptoms (LUTS) as assessed by American Urologic Association (AUA) urinary symptom score > than 8, (suggestive of moderate LUTS) prostate size > 40cc, no prostate nodule/tenderness/firmness and increased PSA between 4-10ng/ml requiring prostate biopsy will be enrolled. Then, they will have prostate MRIs/needle biopsies and blood/urine collection followed by treatment with Finasteride (standard of care). They will be followed in urology clinic for assessment of LUTS every 6 months and Finasteride responsiveness at the 12-month time point. Prostate biopsy samples will be evaluated for SRD5A2 gene expression/methylation, hormonal androgen/estrogen levels (which will be repeated in blood samples). Prostate MRIs will assess size/inflammatory changes at the start and 3-year time points.
  Interventions: Drug: Finasteride

INTERVENTIONS:
Drug: Finasteride — Patients who are candidates to receive 5ARI therapy, Finasteride, for clinical medical management of lower urinary tract symptoms will begin treatment once deemed eligible. They will be assess every 6 months for changes in urinary symptom scores and their responsiveness to the Finasteride treatment will be assessed at the 12-month time point. MRIs of prostate taken at the start of study and at the 3 year time point will assess prostate size and changes in size as well as degree of inflammatory changes. Gene expression of SRD5A2 as well as methylation pattern will be tested on prostate tissue samples, where hormonal androgen/estrogen levels will also be assessed as they are in blood samples.
  Other Names: Sequential Time Point Study

SUMMARY:
The study is being conducted to learn why some patients with Benign Prostatic Hyperplasia (BPH) do not respond to a commonly used treatment drug, Finasteride. The hope is to find ways to predict which patients will not respond to Finasteride so that, in the future, these patients can be identified prior to offering this treatment and they can be offered alternative treatment strategies in its place. The aim is to see if noninvasive techniques such as MRI can detect inflammation of the prostate to assist with early detection of those who will and who will not respond to Finasteride.

DETAILED DESCRIPTION:
Over 90% of adult males develop lower urinary tract symptoms (LUTS) secondary to bladder outlet obstruction by age 80, rendering benign prostatic hyperplasia (BPH) the most common proliferative abnormality in humans. LUTS secondary to BPH negatively impact the quality of life of 210 million men globally, accounting for significant life years lost, in addition to costing the US healthcare system over $4 billion per year. Medical therapy for the management of BPH, which includes α-adrenergic blockers (e.g., doxazosin, terazosin, tamsulosin or alfuzosin) and 5α reductase inhibitors (5ARI, i.e., finasteride or dutasteride) targets both stromal and epithelial cells in the prostate gland. Utilization of 5ARI remains ineffective in many patients, leading to invasive therapies in many patients. 5ARI's are the only class of BPH-related drugs that reduce prostate size for the alleviation of LUTS. However, the Medical Therapy of Prostatic Symptoms (MTOPS) trial, which randomized 3047 men, showed that 34% of BPH patients did not respond to individualized treatment with finasteride or doxazosin, while combining the 5ARI and α-blocker relieved LUTS in 66% of BPH patients. Resistance to 5ARI therapy is a major factor limiting the effectiveness of these agents in the management of BPH. Therefore, understanding the molecular pathogenesis of 5ARI resistance is a High-Priority Recommendation of the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) Prostate Research Strategic Plan. However, it is not yet possible to predict responders vs. non-responders to 5ARI therapy, which creates a significant gap in our ability to effectively manage patients with BPH.

5α reductase (5-AR) plays a critical role in the normal development of the human prostate and in the pathogenesis and progression of prostatic diseases. There are three types of 5-AR isozymes, Steroid 5 Alpha-Reductase 1, 2 3 (SRD5A1, SRD5A2 and SRD5A3), which are encoded by three distinct corresponding genes, SRD5A1, SRD5A2 and SRD5A3. Many studies suggest that all three 5-AR enzymes are expressed in prostate tissues; however, SRD5A2 is the predominant enzyme responsible for prostate development and growth. In addition, since the most commonly prescribed 5ARI, finasteride, is an inhibitor of SRD5A2, regulation of SRD5A2 will remain the focus of this study.

It was previously shown that the mechanism of somatic suppression of SRD5A2 during adulthood is dependent on epigenetic changes in the promoter region of the SRD5A2 gene. DNA methylation is one of the most common epigenetic mechanisms affecting gene expression. Methylation of Cytosine-Phosphate-Guanine (CpG) islands has been associated with the regulation of genes during development, cancer initiation, and metastasis. Since the prostate is the only solid organ that grows during adulthood as a result of androgen exposure, it can be considered a benign tumor growth throughout adulthood. Therefore, similar to the neoplastic initiation and progression of many cancers, including prostate cancer, epigenetic changes and variable expression of SRD5A2 in benign prostate tissue is a plausible molecular mechanism.

Finasteride, the most commonly prescribed 5ARI, is an inhibitor of SRD5A2. Finasteride has been shown in several large clinical trials to reduce prostate size by 20%, improve urinary flow rate, and improve urinary bothersome symptom scores in men suffering from bladder outlet obstruction caused by BPH. Despite their widespread use and clinical effectiveness, 25% to 30% of patients are resistant to the therapeutic effects of 5ARIs and another 5% to 7% of patients develop worsening symptoms and ultimately may require surgery. Given their age and comorbidities, these patients are often not ideal candidates for surgery. Therefore, understanding the mechanisms of 5ARI treatment failure may pave the way for the development of new medical therapies appropriately targeted to these specific patient groups and is a desirable way to move forward with precision medicine. This proposed work is based on the premise that epigenetic changes to SRD5A2 account for the significant number of patients who are unresponsive to 5ARI therapy. The goal is to assess SRD5A2 methylation and expression as a gene signature to predict which patients will respond to 5ARI therapy.

The information gained from this proposal will pave the way toward the development of predictive biomarker assays that can be used to evaluate resistance to BPH-related therapies and allow clinicians to select alternate therapies for managing the most common proliferative disorder affecting men worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Male (physiological);
* Age ≥ 50;
* Eligible for treatment with 5ARI therapy;
* Presence of lower urinary tract symptoms secondary to BPH;
* Prostate size >40cc by digital rectal examination;
* Absence of prostate nodule, tenderness or firmness;
* Mildly elevated PSA's >1.5 ng/ml and ≤ 40 ng/ml;
* Undergoing clinically indicated prostate biopsy for elevated prostate-specific antigen (PSA).

Exclusion Criteria:

* Diagnosis of any prostatic malignancy or precancerous lesions (atypical glandular foci and prostatic intraepithelial neoplasia);
* Treatment with 5ARI (Finasteride or Dutasteride) within six months of study enrollment;
* Current urinary tract infection;
* Previous pelvic radiation;
* Previous treatment with demethylating drugs;
* Diagnosis of multiple sclerosis, Alzheimer's, Parkinson's, neurological deficits in the judgment of the investigator;
* Unable or unwilling to undergo MRI due to implants, claustrophobia, etc.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostatic disease are limited to biologically male individuals.
Enrollment: 120 (Estimated)
Dates: Start 2020-09-25 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Finasteride treatment effect on lower urinary tract symptom improvement by urinary symptom score | Assessment of Finasteride responsiveness through changes in urinary symptoms will be completed at 6 month intervals during clinic visits, and treatment efficacy will be determined after the first 12 months.
  Validated questions of the AUA Urinary Symptom Score will be used every 6 months to assess efficacy of Finasteride treatment in improving lower urinary tract symptoms in the patient population. Based on previous randomized trials, it will be determined whether the patient is responsive or resistant to the treatment dependent on changes in their AUA Urinary Symptom Score at the first 12 month mark. For patients who are resistant to Finasteride, other medical or surgical treatments will be offered, and the patients will be removed from the study.

CONTACTS AND LOCATIONS:
Overall Officials: Aria F. Olumi, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Vos T, Flaxman AD, Naghavi M, Lozano R, Michaud C, Ezzati M, Shibuya K, Salomon JA, Abdalla S, Aboyans V, Abraham J, Ackerman I, Aggarwal R, Ahn SY, Ali MK, Alvarado M, Anderson HR, Anderson LM, Andrews KG, Atkinson C, Baddour LM, Bahalim AN, Barker-Collo S, Barrero LH, Bartels DH, Basanez MG, Baxter A, Bell ML, Benjamin EJ, Bennett D, Bernabe E, Bhalla K, Bhandari B, Bikbov B, Bin Abdulhak A, Birbeck G, Black JA, Blencowe H, Blore JD, Blyth F, Bolliger I, Bonaventure A, Boufous S, Bourne R, Boussinesq M, Braithwaite T, Brayne C, Bridgett L, Brooker S, Brooks P, Brugha TS, Bryan-Hancock C, Bucello C, Buchbinder R, Buckle G, Budke CM, Burch M, Burney P, Burstein R, Calabria B, Campbell B, Canter CE, Carabin H, Carapetis J, Carmona L, Cella C, Charlson F, Chen H, Cheng AT, Chou D, Chugh SS, Coffeng LE, Colan SD, Colquhoun S, Colson KE, Condon J, Connor MD, Cooper LT, Corriere M, Cortinovis M, de Vaccaro KC, Couser W, Cowie BC, Criqui MH, Cross M, Dabhadkar KC, Dahiya M, Dahodwala N, Damsere-Derry J, Danaei G, Davis A, De Leo D, Degenhardt L, Dellavalle R, Delossantos A, Denenberg J, Derrett S, Des Jarlais DC, Dharmaratne SD, Dherani M, Diaz-Torne C, Dolk H, Dorsey ER, Driscoll T, Duber H, Ebel B, Edmond K, Elbaz A, Ali SE, Erskine H, Erwin PJ, Espindola P, Ewoigbokhan SE, Farzadfar F, Feigin V, Felson DT, Ferrari A, Ferri CP, Fevre EM, Finucane MM, Flaxman S, Flood L, Foreman K, Forouzanfar MH, Fowkes FG, Franklin R, Fransen M, Freeman MK, Gabbe BJ, Gabriel SE, Gakidou E, Ganatra HA, Garcia B, Gaspari F, Gillum RF, Gmel G, Gosselin R, Grainger R, Groeger J, Guillemin F, Gunnell D, Gupta R, Haagsma J, Hagan H, Halasa YA, Hall W, Haring D, Haro JM, Harrison JE, Havmoeller R, Hay RJ, Higashi H, Hill C, Hoen B, Hoffman H, Hotez PJ, Hoy D, Huang JJ, Ibeanusi SE, Jacobsen KH, James SL, Jarvis D, Jasrasaria R, Jayaraman S, Johns N, Jonas JB, Karthikeyan G, Kassebaum N, Kawakami N, Keren A, Khoo JP, King CH, Knowlton LM, Kobusingye O, Koranteng A, Krishnamurthi R, Lalloo R, Laslett LL, Lathlean T, Leasher JL, Lee YY, Leigh J, Lim SS, Limb E, Lin JK, Lipnick M, Lipshultz SE, Liu W, Loane M, Ohno SL, Lyons R, Ma J, Mabweijano J, MacIntyre MF, Malekzadeh R, Mallinger L, Manivannan S, Marcenes W, March L, Margolis DJ, Marks GB, Marks R, Matsumori A, Matzopoulos R, Mayosi BM, McAnulty JH, McDermott MM, McGill N, McGrath J, Medina-Mora ME, Meltzer M, Mensah GA, Merriman TR, Meyer AC, Miglioli V, Miller M, Miller TR, Mitchell PB, Mocumbi AO, Moffitt TE, Mokdad AA, Monasta L, Montico M, Moradi-Lakeh M, Moran A, Morawska L, Mori R, Murdoch ME, Mwaniki MK, Naidoo K, Nair MN, Naldi L, Narayan KM, Nelson PK, Nelson RG, Nevitt MC, Newton CR, Nolte S, Norman P, Norman R, O'Donnell M, O'Hanlon S, Olives C, Omer SB, Ortblad K, Osborne R, Ozgediz D, Page A, Pahari B, Pandian JD, Rivero AP, Patten SB, Pearce N, Padilla RP, Perez-Ruiz F, Perico N, Pesudovs K, Phillips D, Phillips MR, Pierce K, Pion S, Polanczyk GV, Polinder S, Pope CA 3rd, Popova S, Porrini E, Pourmalek F, Prince M, Pullan RL, Ramaiah KD, Ranganathan D, Razavi H, Regan M, Rehm JT, Rein DB, Remuzzi G, Richardson K, Rivara FP, Roberts T, Robinson C, De Leon FR, Ronfani L, Room R, Rosenfeld LC, Rushton L, Sacco RL, Saha S, Sampson U, Sanchez-Riera L, Sanman E, Schwebel DC, Scott JG, Segui-Gomez M, Shahraz S, Shepard DS, Shin H, Shivakoti R, Singh D, Singh GM, Singh JA, Singleton J, Sleet DA, Sliwa K, Smith E, Smith JL, Stapelberg NJ, Steer A, Steiner T, Stolk WA, Stovner LJ, Sudfeld C, Syed S, Tamburlini G, Tavakkoli M, Taylor HR, Taylor JA, Taylor WJ, Thomas B, Thomson WM, Thurston GD, Tleyjeh IM, Tonelli M, Towbin JA, Truelsen T, Tsilimbaris MK, Ubeda C, Undurraga EA, van der Werf MJ, van Os J, Vavilala MS, Venketasubramanian N, Wang M, Wang W, Watt K, Weatherall DJ, Weinstock MA, Weintraub R, Weisskopf MG, Weissman MM, White RA, Whiteford H, Wiersma ST, Wilkinson JD, Williams HC, Williams SR, Witt E, Wolfe F, Woolf AD, Wulf S, Yeh PH, Zaidi AK, Zheng ZJ, Zonies D, Lopez AD, Murray CJ, AlMazroa MA, Memish ZA. Years lived with disability (YLDs) for 1160 sequelae of 289 diseases and injuries 1990-2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2163-96. doi: 10.1016/S0140-6736(12)61729-2. PMID 23245607
- [Background] Saigal CS, Joyce G. Economic costs of benign prostatic hyperplasia in the private sector. J Urol. 2005 Apr;173(4):1309-13. doi: 10.1097/01.ju.0000152318.79184.6f. PMID 15758787
- [Background] Chapple CR. Pharmacological therapy of benign prostatic hyperplasia/lower urinary tract symptoms: an overview for the practising clinician. BJU Int. 2004 Sep;94(5):738-44. doi: 10.1111/j.1464-410X.2004.05022.x. PMID 15329091
- [Background] Sarma AV, Jacobson DJ, McGree ME, Roberts RO, Lieber MM, Jacobsen SJ. A population based study of incidence and treatment of benign prostatic hyperplasia among residents of Olmsted County, Minnesota: 1987 to 1997. J Urol. 2005 Jun;173(6):2048-53. doi: 10.1097/01.ju.0000158443.13918.d6. PMID 15879823
- [Background] McConnell JD, Bruskewitz R, Walsh P, Andriole G, Lieber M, Holtgrewe HL, Albertsen P, Roehrborn CG, Nickel JC, Wang DZ, Taylor AM, Waldstreicher J. The effect of finasteride on the risk of acute urinary retention and the need for surgical treatment among men with benign prostatic hyperplasia. Finasteride Long-Term Efficacy and Safety Study Group. N Engl J Med. 1998 Feb 26;338(9):557-63. doi: 10.1056/NEJM199802263380901. PMID 9475762
- [Background] McConnell JD, Roehrborn CG, Bautista OM, Andriole GL Jr, Dixon CM, Kusek JW, Lepor H, McVary KT, Nyberg LM Jr, Clarke HS, Crawford ED, Diokno A, Foley JP, Foster HE, Jacobs SC, Kaplan SA, Kreder KJ, Lieber MM, Lucia MS, Miller GJ, Menon M, Milam DF, Ramsdell JW, Schenkman NS, Slawin KM, Smith JA; Medical Therapy of Prostatic Symptoms (MTOPS) Research Group. The long-term effect of doxazosin, finasteride, and combination therapy on the clinical progression of benign prostatic hyperplasia. N Engl J Med. 2003 Dec 18;349(25):2387-98. doi: 10.1056/NEJMoa030656. PMID 14681504
- [Background] Roehrborn CG, Oyarzabal Perez I, Roos EP, Calomfirescu N, Brotherton B, Wang F, Palacios JM, Vasylyev A, Manyak MJ. Efficacy and safety of a fixed-dose combination of dutasteride and tamsulosin treatment (Duodart((R)) ) compared with watchful waiting with initiation of tamsulosin therapy if symptoms do not improve, both provided with lifestyle advice, in the management of treatment-naive men with moderately symptomatic benign prostatic hyperplasia: 2-year CONDUCT study results. BJU Int. 2015 Sep;116(3):450-9. doi: 10.1111/bju.13033. Epub 2015 Jan 29. PMID 25565364
- [Background] Bautista OM, Kusek JW, Nyberg LM, McConnell JD, Bain RP, Miller G, Crawford ED, Kaplan SA, Sihelnik SA, Brawer MK, Lepor H. Study design of the Medical Therapy of Prostatic Symptoms (MTOPS) trial. Control Clin Trials. 2003 Apr;24(2):224-43. doi: 10.1016/s0197-2456(02)00263-5. PMID 12689743
- [Background] Kaplan SA, Lee JY, Meehan AG, Kusek JW; MTOPS Research Group. Long-term treatment with finasteride improves clinical progression of benign prostatic hyperplasia in men with an enlarged versus a smaller prostate: data from the MTOPS trial. J Urol. 2011 Apr;185(4):1369-73. doi: 10.1016/j.juro.2010.11.060. Epub 2011 Feb 22. PMID 21334655
- [Background] Wang K, Fan DD, Jin S, Xing NZ, Niu YN. Differential expression of 5-alpha reductase isozymes in the prostate and its clinical implications. Asian J Androl. 2014 Mar-Apr;16(2):274-9. doi: 10.4103/1008-682X.123664. PMID 24457841
- [Background] Imperato-McGinley J, Guerrero L, Gautier T, Peterson RE. Steroid 5alpha-reductase deficiency in man: an inherited form of male pseudohermaphroditism. Science. 1974 Dec 27;186(4170):1213-5. doi: 10.1126/science.186.4170.1213. PMID 4432067
- [Background] Walsh PC, Madden JD, Harrod MJ, Goldstein JL, MacDonald PC, Wilson JD. Familial incomplete male pseudohermaphroditism, type 2. Decreased dihydrotestosterone formation in pseudovaginal perineoscrotal hypospadias. N Engl J Med. 1974 Oct 31;291(18):944-9. doi: 10.1056/NEJM197410312911806. No abstract available. PMID 4413434
- [Background] Livingstone DE, Barat P, Di Rollo EM, Rees GA, Weldin BA, Rog-Zielinska EA, MacFarlane DP, Walker BR, Andrew R. 5alpha-Reductase type 1 deficiency or inhibition predisposes to insulin resistance, hepatic steatosis, and liver fibrosis in rodents. Diabetes. 2015 Feb;64(2):447-58. doi: 10.2337/db14-0249. Epub 2014 Sep 19. PMID 25239636
- [Background] Azzouni F, Godoy A, Li Y, Mohler J. The 5 alpha-reductase isozyme family: a review of basic biology and their role in human diseases. Adv Urol. 2012;2012:530121. doi: 10.1155/2012/530121. Epub 2011 Dec 25. PMID 22235201
- [Background] Stiles AR, Russell DW. SRD5A3: A surprising role in glycosylation. Cell. 2010 Jul 23;142(2):196-8. doi: 10.1016/j.cell.2010.07.003. PMID 20655462
- [Background] Ge R, Wang Z, Bechis SK, Otsetov AG, Hua S, Wu S, Wu CL, Tabatabaei S, Olumi AF. DNA methyl transferase 1 reduces expression of SRD5A2 in the aging adult prostate. Am J Pathol. 2015 Mar;185(3):870-82. doi: 10.1016/j.ajpath.2014.11.020. Epub 2015 Feb 17. PMID 25700986
- [Background] Bechis SK, Otsetov AG, Ge R, Olumi AF. Personalized medicine for the management of benign prostatic hyperplasia. J Urol. 2014 Jul;192(1):16-23. doi: 10.1016/j.juro.2014.01.114. Epub 2014 Feb 25. PMID 24582540
- [Background] Baylin SB, Jones PA. A decade of exploring the cancer epigenome - biological and translational implications. Nat Rev Cancer. 2011 Sep 23;11(10):726-34. doi: 10.1038/nrc3130. PMID 21941284
- [Background] Esteller M. Cancer epigenomics: DNA methylomes and histone-modification maps. Nat Rev Genet. 2007 Apr;8(4):286-98. doi: 10.1038/nrg2005. Epub 2007 Mar 6. PMID 17339880
- [Background] Beltran H, Prandi D, Mosquera JM, Benelli M, Puca L, Cyrta J, Marotz C, Giannopoulou E, Chakravarthi BV, Varambally S, Tomlins SA, Nanus DM, Tagawa ST, Van Allen EM, Elemento O, Sboner A, Garraway LA, Rubin MA, Demichelis F. Divergent clonal evolution of castration-resistant neuroendocrine prostate cancer. Nat Med. 2016 Mar;22(3):298-305. doi: 10.1038/nm.4045. Epub 2016 Feb 8. PMID 26855148
- [Background] Bechis SK, Otsetov AG, Ge R, Wang Z, Vangel MG, Wu CL, Tabatabaei S, Olumi AF. Age and Obesity Promote Methylation and Suppression of 5alpha-Reductase 2: Implications for Personalized Therapy of Benign Prostatic Hyperplasia. J Urol. 2015 Oct;194(4):1031-7. doi: 10.1016/j.juro.2015.04.079. Epub 2015 Apr 25. PMID 25916673
- [Background] Austin DC, Strand DW, Love HL, Franco OE, Grabowska MM, Miller NL, Hameed O, Clark PE, Matusik RJ, Jin RJ, Hayward SW. NF-kappaB and androgen receptor variant 7 induce expression of SRD5A isoforms and confer 5ARI resistance. Prostate. 2016 Aug;76(11):1004-18. doi: 10.1002/pros.23195. Epub 2016 May 16. PMID 27197599